CLINICAL TRIAL: NCT06789809
Title: Exercise Physiology in Patients With Aortic Aneurysm and Its Correlation With Mechanical Properties of Aortic Tissue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Deborah Kwon, MD, Principal Investigator, The Cleveland Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-310
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Controls (Experimental): Exercise MRI
  Interventions: Diagnostic Test: Exercise MRI
- Aneurysm Being Monitored (Experimental): Exercise MRI
  Interventions: Diagnostic Test: Exercise MRI
- Pre-operative Aneurysm Patients (Experimental): Exercise MRI
  Interventions: Diagnostic Test: Exercise MRI

INTERVENTIONS:
Diagnostic Test: Exercise MRI — Exercise stress MRI with ergometer

SUMMARY:
Aortic aneurysm patients benefit from exercise yet patients and physicians do not know a safe level. Cardiac MRI (CMR) is the most comprehensive imaging modality for phenotypic evaluation of patients with cardiac disease but it has not been used to study aneurysm patients. The purpose of this project is use exercise CMR to understand regional aortic function and quantify aortic elasticity in these populations while exercising. This project will correlate the exercise CMR data with the biomechanical properties of the patient's aortic tissue, including epiaortic ultrasound and TEE performed during aortic repair, and explanted aortic specimens subjected to ex vivo uniaxial tensile testing. Correlating this data with aortic response to exercise will allow us to understand how aortic size, in vivo circumferential strain values, ex vivo aortic efficiency and mechanical failure all relate to exercise physiology.

DETAILED DESCRIPTION:
Engaging in regular exercise in controls lowers blood pressure over time, and this is associated with a lower risk of future aortic complications. However, it is not known what level of exercise is safe for aneurysm patients.

Cardiac MRI (CMR) is the most comprehensive imaging modality for phenotypic evaluation of patients with cardiac disease. It has been limited in its use because exercise stress MRI is not widely available due to the need for MRI safe exercise equipment. However, the Cleveland Clinic has purchased a Lode MRI compatible exercise ergometer that is FDA approved and compatible with our 3T cardiac MRI scanner.

By conducting a study using this imaging modality we will be able to observe aortic blood flow, specifically compliance, distensibility, maximum rates of systolic distension and diastolic recoil, at different locations along the ascending and descending aorta, as well as aortic pulse wave velocity. A more comprehensive analysis of these variables will be critical to understanding how the aorta responds during times of stress in aneurysm patients.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy controls for baseline comparison

   1. Must be 18 years or older
   2. No history of cardiovascular disease, neither hypertension, diabetes nor hypercholesterolemia
2. Aneurysm patients who have not yet been operated on but are currently being monitored

   1. Must be 18 years or older
   2. No history of operation for aortic aneurysm
3. Pre-operative aneurysm patients: imaged pre-operatively and 12 months

   1. Patients admitted at the CCF cardiothoracic services for elective surgery due to aortic aneurysms
   2. Must be 18 years or older

Exclusion Criteria:

For all patients:

* Contra-indication for MRI

  * Heart pacemaker/defibrillator.
  * Electronic/implanted stimulators or devices, including deep brain stimulator, vagus nerve stimulator, bladder stimulator, spine stimulator, neurostimulators; implanted electrodes or wires.
  * Cochlear implant or other ear implants.
  * Implanted drug pumps (insulin, narcotic/pain medications, drugs to treat spasticity).
  * Programmable shunt.
  * Aneurysm clips and coils.
  * Stents (not located in heart).
  * Filters (for example, blood clot filters).
  * Metal fragment in your body or eye (eg, BBs, bullets, shrapnel, metal pieces or shavings).
* Congenital heart diseases such as patent ductus arteriosus, coarctation of aorta, ASD and VSD
* Presence of A-V fistula or intracardiac shunts
* Moderate or severe dysfunction in multiple valves
* Patients with significant claustrophobia
* Patients unable to pedal a supine bicycle
* Those who require supplemental oxygen

Specific Exclusion Criteria:

1. Healthy controls for baseline comparison

   1. Excluded if using cardioprotective medication
   2. Have a bicuspid aortic valve diagnosed using MRI
2. Pre-operative aneurysm patients: imaged pre-operatively and at 12 months a. Patients with traumatic aortic rupture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Arterial Compliance | up to 12 months
  Absolute change in arterial volume for a change in pressure

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Kwon, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No